CLINICAL TRIAL: NCT02744326
Title: Improving Outcomes for Youth Visiting the Emergency Department With Mental Health Issues
Brief Title: Outcomes in Youth Visiting the ED With Mental Health Issues: a Pilot Text Based Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1603-026
Record Dates: First submitted 2016-04-14; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Mental Health Disorder; Mental and Behavioral Disorder; Self-inflicted Injury
MeSH Terms: conditions — Mental Disorders; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text message reminder group (Experimental): A subset of patients discharged from the ED with an outpatient referral will be randomized to receive text message reminders to attend or schedule a follow-up outpatient referral.
  Interventions: Behavioral: Text message reminders
- Usual Care group (No Intervention): A subset of patients discharged from the ED with an outpatient referral will be randomized to receive the usual standard of care.

INTERVENTIONS:
Behavioral: Text message reminders — Patients assigned to the intervention group will receive a series of 7 to 10 text message reminders to schedule or attend their follow-up appointment.
  Arms: Text message reminder group

SUMMARY:
The investigators will conduct a prospective study and a randomized controlled trial (RCT) involving children and adolescents presenting with a primary mental health (MH) concern to the emergency departments (EDs) of Children's Hospitals and Clinics of Minnesota (CH). The investigators will characterize the primary MH concerns of 800 patients and assess their baseline access to and utilization of external resources. All enrolled patients will be followed 3-months after their initial visit to determine ED revisits and identify factors associated with connection to outpatient care. The RCT portion of the study will involve 200 patients discharged from the ED with a referral to an outpatient MH provider, and will test a novel text-message communication method by which parents/caregivers can be encouraged to complete follow-up care for their child. The experimental group will receive tailored text message reminders regarding follow-up appointments.

Relevance: Pediatric ED visits for MH issues are increasing, but the current system of managing these patients is not optimal. More information is needed to accelerate change and to efficiently invest in improving services available to MH patients. Specifically, information is needed on which MH populations need to be targeted, and on simple, reproducible interventions which improve connection with community resources. The proposed study will collect vital information needed to develop programs that improve outcomes and reduce ED revisits in pediatric patients visiting the EDs at CH with primary MH concerns, and will set the stage for future work focused on improving core and outcomes for MH youth.

DETAILED DESCRIPTION:
Background/Significance The number of youth visiting the ED with MH issues has risen dramatically in the last decade.1 EDs have become a safety net for a strained mental health system that is under resourced and lacks adequate services to meet demands at the impatient and outpatient level.2 EDs bear a high burden of caring for children and adolescents with acute psychiatric illness, and pediatric patients with MH-related visits require substantial ED resources.2,3 Visits to the ED for MH are longer, more likely to be triaged to urgent evaluation and result in more admissions or transfers compared to visits for other reasons.4,5 ED revisits are also are also common in pediatric MH patients, with a recent study finding return rates of 6-9% within 72 hours, and return rates around 30% over a 4-year study period.6 ED visits for children and adolescents with MH concerns are resource intensive, and further research will be crucial for improving the management of these patients.2,3

Information lacking on resources needed by MH diagnostic subgroup:

MH issues encountered by ED physicians cover a broad range of diagnoses. Bardach et al. examined MH hospitalizations and identified the following as the most common diagnostic subgroups: depression, bipolar disorder, psychosis, externalizing disorder, anxiety disorder, ADHD, eating disorder, substance abuse, reaction disorder and autism.7 ED visits for MH concerns are often thought to mainly involve suicide attempts, self-harm behavior or psychosis, but a recent study of a large urban pediatric ED found that almost half of the visits were for behavioral problems.8 Preliminary data has described that almost half of the behavioral assessments done at CH in 2013 were on individuals with developmental disorders (i.e. autism spectrum disorders). The number of MH ED visits for behavioral issues is growing, but there is limited information regarding this population.8 Overall, the ED experience has not been well documented based upon diagnostic subgroup, but there are critical differences in MH patients depending on their primary concern, specifically connection to outpatient resources and risk of ED revisit.8,9 In order to more efficiently help MH youth it is crucial to obtain information regarding services, and how this differs by diagnostic subgroup.8

Text-messaging to improve MH referral follow-up:

The ED represents a suboptimal care setting for MH youth but does provide an important opportunity to identify children and adolescents in crisis and connect them with external resources.8 Unfortunately, successful follow-up with MH resources by ED patients has been shown to be low, with some studies finding follow-up rates below 30%.10,11 A recent study found that 66% of patients visiting the ED with suicidal behaviors successfully followed up with a mental health provider, a more positive number, but one that still shows a large need for improvement.12 Strategies are needed to improve successful follow-up with MH outpatient referrals as failure to comply with ED discharge guidelines could result in worsening of symptoms and return visits to the ED. While ED providers have a unique opportunity to identify MH youth and provide referrals, they also have limited time and resources. If an intervention is to be incorporated into usual care in the ED, it must be simple, efficient, and easy to replicate. Automated text messaging reminders have been shown to increase attendance to healthcare appointments.13 Over 90% of Americans reported owning a cell phone in 2013, and 81% report using their cell phone to send or receive text messages.14 In addition, the cost and personnel requirements needed to implement an automated text message based system are low, making this a unique intervention technique that could be easily incorporated into usual care in any ED.15 A recent study found that automated text message appointment reminders improved follow-up attendance to primary or specialty care in adult ED patients.15 Additional research is needed to examine the potential of a text message strategy to increase attendance to follow-up appointments in a diverse population of youth visiting the ED the MH concerns.

Conclusion:

The overall goal of the proposed study is to collect vital information needed to develop programs that improve outcomes and reduce revisits in children and adolescents who present to the ED with primary MH concerns. Pediatric ED visits for MH issues are increasing.1 The current system is in need of improvement, yet more information is needed to accelerate change, including information on which MH populations need to be targeted, and on simple, reproducible interventions which improve connection with community resources. The proposed project will collect data on a cohort of MH patients from two large urban EDs to characterize diagnostic subgroups and current access to care, will follow all patients 3-months post visit to identify risk factors for ED revisits and barriers to outpatient care, and will test a novel text message reminder system focused on improving the linkage of MH patients with follow-up referrals. The EDs of CH provide the vast majority of emergent pediatric care within the Twin City Metro area, and a substantial proportion of these visits are mental health related. The proposed project provides a unique opportunity to meet the study goals, and sets the stage for future work focused on improving care and outcomes for MH youth.

Research Question

1. Which pediatric MH patients visiting the ED at CH are in the most need of additional support (lowest baseline access to and utilization of outpatient care, highest risk of ED revisit, lowest follow-up with outpatient referrals)?
2. Does a targeted text-message communication method improve compliance with ED discharge in pediatric MH patients?

Specific Aims and Hypotheses

1. Characterize the primary MH concerns of children and adolescent visiting the EDs of CH and assesses their baseline access to and utilization of external MH resources.

   Hypothesis: MH patients will represent several subgroups of primary concerns and these subgroups will differ in their baseline connection to and utilization of community resources.
2. Follow all enrolled MH patients post visit to determine factors associated with ED revisits and barriers to outpatient care.

   Hypothesis: Patients who have public or no insurance, who visit the ED with self-inflicted injuries, or who identify multiple barriers to connecting with outpatient MH care will have higher rates of ED revisits.
3. Develop and test a novel text-message communication method focused on increasing rates of discharge referral follow-up in ED patients with MH concerns.

Hypothesis: Patients randomized to a text-message communication system will have higher rates of follow-up care and lower rates of ED revisit compared to patients who receive usual care

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17.999 years
* Assessed by social work in the ED for mental health concern
* Parent present and able to consent
* Phone able to receive text messages (for RCT portion only)

Exclusion Criteria:

* Non-English Speaking parents
* Medical condition preventing enrollment, such as a condition which requires immediated hospital procedures or admission
* Suspected abuse

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Outpatient care post Emergency Department Visit | 3 months
  Did the patient attend follow-up outpatient care visit(s) after visiting the ED

SECONDARY OUTCOMES:
Emergency Department return visit | 3 months
  Did the patient return to the Emergency Department for a mental health related reason, in the 3 months following the initial visit.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Cutler, PhD, Principal Investigator — Children's Hospitals and Clinics of Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simon AE, Schoendorf KC. Emergency department visits for mental health conditions among US children, 2001-2011. Clin Pediatr (Phila). 2014 Dec;53(14):1359-66. doi: 10.1177/0009922814541806. Epub 2014 Jul 7. PMID 25006117
- [Background] Dolan MA, Fein JA; Committee on Pediatric Emergency Medicine. Pediatric and adolescent mental health emergencies in the emergency medical services system. Pediatrics. 2011 May;127(5):e1356-66. doi: 10.1542/peds.2011-0522. Epub 2011 Apr 25. PMID 21518712
- [Background] Grupp-Phelan J, Mahajan P, Foltin GL, Jacobs E, Tunik M, Sonnett M, Miller S, Dayan P; Pediatric Emergency Care Applied Research Network. Referral and resource use patterns for psychiatric-related visits to pediatric emergency departments. Pediatr Emerg Care. 2009 Apr;25(4):217-20. doi: 10.1097/pec.0b013e31819e3523. PMID 19382317
- [Background] Case SD, Case BG, Olfson M, Linakis JG, Laska EM. Length of stay of pediatric mental health emergency department visits in the United States. J Am Acad Child Adolesc Psychiatry. 2011 Nov;50(11):1110-9. doi: 10.1016/j.jaac.2011.08.011. Epub 2011 Oct 2. PMID 22023999
- [Background] Mahajan P, Alpern ER, Grupp-Phelan J, Chamberlain J, Dong L, Holubkov R, Jacobs E, Stanley R, Tunik M, Sonnett M, Miller S, Foltin GL; Pediatric Emergency Care Applied Research Network (PECARN). Epidemiology of psychiatric-related visits to emergency departments in a multicenter collaborative research pediatric network. Pediatr Emerg Care. 2009 Nov;25(11):715-20. doi: 10.1097/PEC.0b013e3181bec82f. PMID 19864967
- [Background] Newton AS, Ali S, Johnson DW, Haines C, Rosychuk RJ, Keaschuk RA, Jacobs P, Cappelli M, Klassen TP. Who comes back? Characteristics and predictors of return to emergency department services for pediatric mental health care. Acad Emerg Med. 2010 Feb;17(2):177-86. doi: 10.1111/j.1553-2712.2009.00633.x. PMID 20370747
- [Background] Bardach NS, Coker TR, Zima BT, Murphy JM, Knapp P, Richardson LP, Edwall G, Mangione-Smith R. Common and costly hospitalizations for pediatric mental health disorders. Pediatrics. 2014 Apr;133(4):602-9. doi: 10.1542/peds.2013-3165. Epub 2014 Mar 17. PMID 24639270
- [Background] Frosch E, McCulloch J, Yoon Y, DosReis S. Pediatric emergency consultations: prior mental health service use in suicide attempters. J Behav Health Serv Res. 2011 Jan;38(1):68-79. doi: 10.1007/s11414-009-9192-0. Epub 2009 Sep 19. PMID 19768551
- [Background] Smith MW, Stocks C, Santora PB. Hospital readmission rates and emergency department visits for mental health and substance abuse conditions. Community Ment Health J. 2015 Feb;51(2):190-7. doi: 10.1007/s10597-014-9784-x. Epub 2015 Jan 7. PMID 25563483
- [Background] Grupp-Phelan J, McGuire L, Husky MM, Olfson M. A randomized controlled trial to engage in care of adolescent emergency department patients with mental health problems that increase suicide risk. Pediatr Emerg Care. 2012 Dec;28(12):1263-8. doi: 10.1097/PEC.0b013e3182767ac8. PMID 23187979
- [Background] Sobolewski B, Richey L, Kowatch RA, Grupp-Phelan J. Mental health follow-up among adolescents with suicidal behaviors after emergency department discharge. Arch Suicide Res. 2013;17(4):323-34. doi: 10.1080/13811118.2013.801807. PMID 24224667
- [Background] Gurol-Urganci I, de Jongh T, Vodopivec-Jamsek V, Atun R, Car J. Mobile phone messaging reminders for attendance at healthcare appointments. Cochrane Database Syst Rev. 2013 Dec 5;2013(12):CD007458. doi: 10.1002/14651858.CD007458.pub3. PMID 24310741
- [Background] Arora S, Burner E, Terp S, Nok Lam C, Nercisian A, Bhatt V, Menchine M. Improving attendance at post-emergency department follow-up via automated text message appointment reminders: a randomized controlled trial. Acad Emerg Med. 2015 Jan;22(1):31-7. doi: 10.1111/acem.12503. Epub 2014 Nov 11. PMID 25388481